CLINICAL TRIAL: NCT00425438
Title: A Randomized, Open-label Study to Compare the Effect of CellCept Plus Corticosteroids, and Cyclophosphamide Plus Corticosteroids Followed by Azathioprine, on Remission Rate in Patients With Lupus Nephritis
Brief Title: A Study of CellCept (Mycophenolate Mofetil) in Patients With Lupus Nephritis.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early for administrative reasons.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19978
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Adrenal Cortex Hormones; Prednisolone; Azathioprine; Cyclophosphamide

ARMS (2):
- Mycophenolate Mofetil (Experimental): Participants received mycophenolate mofetil (MMF) 0.5 grams (g), orally (PO), twice daily (BID) from Day 0 to the end of Week 1, followed by 1.0 g, PO, BID from Weeks 2 through 24, and 0.75 g, PO, BID from Weeks 32 to 48. Participants also received prednisolone 0.75 to 1.0 milligrams per kilogram (mg/kg), PO, once per day, up to a maximum of 60 mg per day from Weeks 1 through 4, reduced by 10 mg per day every 2 weeks until dose reaches 40 mg per day, followed by a reduction of 5 mg per day every 2 weeks until dose reaches 10 mg per day up to Week 48.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Corticosteroids
- Cyclophosphamide/Azathioprine (Active Comparator): Participants received cyclophosphamide 0.75 grams per square meter (g/m^2), intravenously (IV), every 4 weeks from Weeks 1 through 4, and 0.5 to (-) 1.0 g/m^2, IV, to maintain a minimum white blood cell (WBC) count of greater than or equal to (≥) 2500 per cubic millimeter (mm^3) every 4 weeks from Weeks 5 through 24. Participants also received azathioprine 100 mg, PO, daily for participants with a body weight of 50 to 70 kg and 150 mg, PO, daily for subjects with a body weight of more than 70 kg from Weeks 25 through 48. Participants also received prednisolone 0.75 to 1.0 mg/kg, PO, once per day, up to a maximum of 60 mg per day from Weeks 1 through 4, reduced by 10 mg per day every 2 weeks until dose reaches 40 mg per day, followed by a reduction of 5 mg per day every 2 weeks until dose reaches 10 mg per day up to Week 48.
  Interventions: Drug: Corticosteroids; Drug: Azathioprine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 0.5 g PO BID from Day 0 to the end of Week 1, followed by 1.0 g PO BID from Weeks 2 through 24, and 0.75 g PO BID from Weeks 32 to 48
  Other Names: CellCept
  Arms: Mycophenolate Mofetil
Drug: Corticosteroids — 0.75 to 1.0 mg/kg/d PO (up to 60 kg/day) from Weeks 1 through 4; reduced by 10 mg/day every 2 weeks until dose reaches 40 mg/day, followed by a reduction of 5 mg/day every 2 weeks until dose reaches 10 mg/day up to Week 48
  Other Names: Prednisolone
Drug: Azathioprine — 100 mg PO daily for participants with a body weight of 50 to 70 kg,150 mg PO daily for subjects with a body weight of more than 70 kg up to Week 48
  Arms: Cyclophosphamide/Azathioprine
Drug: Cyclophosphamide — 0.75 g/m^2 IV every 4 weeks from Weeks 1 through 4, and 0.5-1.0 g/m^2 to maintain a minimum WBC count of ≥ 2500 per mm^3 from Weeks 5 through 24
  Arms: Cyclophosphamide/Azathioprine

SUMMARY:
This 2 arm study will compare the efficacy and safety of CellCept plus corticosteroids, versus cyclophosphamide plus corticosteroids in the induction phase followed by azathioprine in the maintenance phase, in maintaining remission and renal function in patients with lupus nephritis. Patients will be randomized to receive CellCept 1g bid po plus corticosteroids for 24 weeks, followed by CellCept 0.75g bid po plus corticosteroids for the following 24 weeks, or cyclophosphamide 0.5-1.0g/m2 monthly plus corticosteroids for 24 weeks, followed by azathioprine 2mg/kg/day po plus corticosteroids for the following 24 weeks. Response rate will be assessed at the end of the induction phase, and at the end of study. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* systemic lupus erythematosus;
* histological diagnosis of lupus nephritis.

Exclusion Criteria:

* not in need of immunosuppressive treatment (in addition to corticosteroids);
* continuous dialysis starting >2 weeks before randomization, with an anticipated duration of >8 weeks;
* previous or planned kidney transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- China (6):
  - Beijing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Shenyang

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil: Participants received mycophenolate mofetil (MMF) 0.5 grams (g), orally (PO), twice daily (BID) from Day 0 to the end of Week 1, followed by 1.0 g, PO, BID from Weeks 2 through 24, and 0.75 g, PO, BID up to 48 weeks after Week 24. Participants also received prednisolone 0.75 to 1.0 milligrams per kilogram (mg/kg), PO, once per day, up to a maximum of 60 mg per day from Weeks 1 through 4, reduced by 10 mg per day every 2 weeks until dose reached 40 mg/day, followed by a reduction of 5 mg/day every 2 weeks until dose reached 10 mg per day up to Week 48.
- Cyclophosphamide, Azathioprine: Participants received cyclophosphamide 0.75 grams per square meter (g/m^2), intravenously (IV), every 4 weeks from Weeks 1 through 4, and 0.5 to (-) 1.0 g/m^2, IV, to maintain a minimum white blood cell (WBC) count of greater than or equal to (≥) 2500 per cubic millimeter (/mm^3) every 4 weeks from Weeks 5 through 24. Participants also received azathioprine 100 mg, PO, daily for participants with a body weight of 50 to 70 kg and 150 mg, PO, daily for participants with a body weight of more than 70 kg from Weeks 25 through 48. Participants also received prednisolone 0.75 to 1.0 mg/kg, PO, once per day, up to a maximum of 60 mg per day from Weeks 1 through 4, reduced by 10 mg per day every 2 weeks until dose reached 40 mg/day, followed by a reduction of 5 mg/day every 2 weeks until dose reached 10 mg per day up to Week 48.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Started | 25 | 27
Completed | 0 | 0
Not Completed | 25 | 27
Not completed — Termination by Sponsor | 25 | 27

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who recieved at least one dose of study drug.
Groups:
- Cyclophosphamide, Azathioprine: Participants received cyclophosphamide 0.75 g/m^2, IV, every 4 weeks from Weeks 1 through 4, and 0.5-1.0 g/m^2, IV, to maintain a minimum WBC count of 2500/mm^3 every 4 weeks from Weeks 5 through 24. Participants also received azathioprine 100 mg, PO, daily for participants with a body weight of 50 to 70 kg and 150 mg, PO, daily for participants with a body weight of more than 70 kg from Weeks 25 through 48. Participants also received prednisolone 0.75 to 1.0 mg/kg, PO, once per day, up to a maximum of 60 mg per day from Weeks 1 through 4, reduced by 10 mg per day every 2 weeks until dose reached 40 mg/day, followed by a reduction of 5 mg/day every 2 weeks until dose reached 10 mg per day up to Week 48.
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.8) | 31.6 (8.0) | 32.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Secondary Outcome: Complete Response
Description: The median time, in months, to CR was defined as the time from randomization to CR event.
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: Efficacy data were not analyzed because of study termination. The study was terminated early for administrative reasons and no participants completed all planned study visits; therefore efficacy analyses could not be performed.
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Treatment Response Event by End of Treatment
Description: Treatment response was defined by a reduction in the ratio of urine protein to creatinine to <3 mg/mg for participants with nephrotic proteinuria and a decrease of more than 50% in their urine protein to creatinine value from BL for participants with non-nephrotic proteinuria; a stable serum creatinine value or an increase of more than 30% from BL; and having not received IV prednisone after Week 28.
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: as for outcome 1
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With a Decrease of 25% or 50% in Glomerular Filtration Rate (GFR)
Description: GFR was calculated according to the simplified modification of diet in renal disease (MDRD) formula.
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: as for outcome 1
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Terminating Treatment
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: as for outcome 1
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Treatment failure was defined as the occurrence of any of the following: death; chronic renal failure requiring dialysis or kidney transplantation; an increase in average serum creatinine values by 2-fold for 2 consecutive measures from BL, and a increase by 2-fold for 2 consecutive measures in at least 4 weeks; recurrent kidney disease defined by, proteinuria, a doubling in the ratio of urine protein to creatinine from BL and a urinary protein value of <0.5 g/24h or greater than (>) 1 g/24h or >0.5 g/24h or >2 g/24h at Week 24, kidney disease, defined by an increase in serum creatinine of 25% from BL along with a doubling of urinary protein of at least 2 g/24h, and hematuria, 2 or more blood cells per urine dipstick test.
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: as for outcome 1
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Complete Response (CR) by the End of Treatment - Percentage of Participants With an Event
Description: CR was defined as a urinary protein value of less than (<) 500 mg per 24 hours (mg/24h) and no hematuria or cellular casts in the urine, and a stable serum creatinine value within the range of plus or minus (±) 25 percent (%) of baseline (BL) or some improvement.
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: as for outcome 1
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening, Day 0, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48.
Description: All participants who received at least 1 dose of study treatment were included in the safety analysis population.
Arm/Group | Mycophenolate Mofetil | Cyclophosphamide, Azathioprine
Serious Adverse Events (participants affected / at risk) | 8/25 | 5/27
Other Adverse Events (participants affected / at risk) | 13/25 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil (N=25) | Cyclophosphamide, Azathioprine (N=27)
Lung infection (Infections and infestations) | 1 | 2
Pyrexia (General disorders) | 1 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Acute renal failure (Renal and urinary disorders) | 1 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0
Hospitalization (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil (N=25) | Cyclophosphamide, Azathioprine (N=27)
Oedema peripheral (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4
Dyschezia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum decreased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Eyelid oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.